CLINICAL TRIAL: NCT02945085
Title: 3D Team Care for Cognitively Vulnerable Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Connecticut (Other)
Responsible Party: Principal Investigator, Fortinsky, Richard, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-021-1
Record Dates: First submitted 2016-10-23; First posted 2016-10-26 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Dementia; Depression; Delirium
Keywords: older adults; family caregivers; Medicare Advantage beneficiaries
MeSH Terms: conditions — Dementia; Depression; Delirium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Based Care Team (Experimental): Primarily in-home treatment provided by team led by nurse practitioner with geriatrics and geriatric psychiatry expertise.
  Interventions: Other: Home Based Care Team
- Telephone Based Care Team (Active Comparator): Primarily telephone-based treatment provided by existing care management program offered by collaborating Medicare Advantage insurer.
  Interventions: Other: Telephone Based Care Team

INTERVENTIONS:
Other: Home Based Care Team — Clinical team will conduct comprehensive clinical assessments focused on cognitive impairment and depression, conduct comprehensive medication review and reconciliation, offer Problem Solving Therapy, and offer brief occupational therapy, physical therapy, nutrition, and social support services.
  Arms: Home Based Care Team
Other: Telephone Based Care Team — Telephone contact will be made by nurses. Depending on level of need, follow up telephone and, in some cases, in home visits will be made by nurse or social worker from care management program.
  Arms: Telephone Based Care Team

SUMMARY:
This study addresses how to achieve better outcomes for cognitively vulnerable community-dwelling older adults and their families. Cognitive vulnerability means living with dementia, depression, and/or a recent episode of delirium (the 3Ds). The investigators will test the effectiveness of a team care model focused on the 3Ds (Home Based Care Team) guided by nurse practitioners with expertise in geriatrics and geriatric psychiatry. Specific aims are to determine Home Based Care Team effects on hospitalization or emergency department use, and other outcomes including depression, disability, and quality of life.

DETAILED DESCRIPTION:
This study addresses how to achieve better outcomes for cognitively vulnerable community-dwelling older adults and their families. Cognitive vulnerability means living with dementia, depression, and/or a recent episode of delirium (the 3Ds). Cognitive vulnerability in older adults is often overlooked by primary care and hospital-based providers, and represents a marker for overall vulnerability or frailty often missed when disease-specific approaches are emphasized in the care for older adults. Such patients often cannot adequately self-manage their comorbidities. Many studies of older adults and their families have demonstrated the great burden of living with cognitive vulnerability. The investigators will test the effectiveness of a team care model focused on the 3Ds (Home Based Care Team) guided by nurse practitioners with geriatrics expertise. Other team member disciplines will include pharmacy, social work, occupational and physical therapy, nutrition, and community health worker. Long-term objectives are to determine whether this care model can become a widely available approach for improving healthcare systems for older adults with cognitive vulnerability and their families, while improving outcomes of importance to these patients and families. A project Steering Committee, including cognitively vulnerable patients and family caregivers, will provide extensive input into many aspects of the research process.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of dementia, depression, and/or delirium, based on diagnostic codes found in medical claims data and based on screening at time of study screening.
* Living in the community, including assisted living facility, at time of randomization
* Plan to live in geographic area for 12 months
* Speak or understand English
* Willing to be randomly assigned to intervention or active comparator group

Exclusion Criteria:

* Diagnosed schizophrenia or bipolar disorder
* Bedbound and non-communicative
* Life expectancy <12 months
* Already enrolled in active comparator program
* For individuals with dementia, family caregiver is unavailable or unwilling to enroll in study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 506 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Proportion hospitalized or used emergency department without hospitalization | 12 months
  Evidence of hospitalization or visit to emergency department without hospital admission will be based on data from the Medicare Advantage insurer's medical claims data warehouse.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ9) | 12 months
  This outcome will be used for study participants with depression but not dementia or recent episode of delirium at baseline. Individual scores will be aggregated into group mean scores to compare intervention and active comparator groups on this outcome.
Caregiver Assessment of Function and Upset (CAFU) | 12 months
  This measure yields a score for each individual reflecting level of assistance required to conduct 7 self-care activities of daily living (ADLs) and 8 instrumental ADLs. In a structured interview format, family members report these items for their relatives with dementia and/or a recent history of delirium. Individual scores will be aggregated into group mean scores to compare intervention and active comparator groups on this outcome.
Family caregiver perceived well-being | 12 months
  Self-reported well-being among family caregivers who enroll in the study

OTHER OUTCOMES:
World Health Organization (WHO) Disability Assessment Schedule, 12 item short form. | 12 months
  This measure yields a score for each individual reflecting self-reported degree of difficulty performing physical activities in the home and community. Individual scores will be aggregated into group mean scores to compare intervention and active comparator groups on this outcome.
Quality of Life-Alzheimer's Disease Scale (QOL-AD) | 12 months
  This measure, used with individuals with dementia, yields a score for each individual reflecting self-ratings of poor, fair, good, or excellent on 13 items. Individual scores will be aggregated into group mean scores to compare intervention and active comparator groups on this outcome.
Neuropsychiatric Inventory (NPI-C) | 12 months
  This measure yields a single score that accounts for both frequency and severity of 14 neuropsychiatric symptoms. Family caregivers provide this information in a structured interview format. Individual scores will be aggregated into group mean scores to compare intervention and active comparator groups on this outcome.
Center for Epidemiologic Studies-Depression Scale (CES-D) | 12 months
  This measure will be used to determine severity of depression among family caregivers enrolled in the study.This measure yields a score for each individual reflecting frequency of 20 depression-related symptoms within the previous two weeks. Individual scores will be aggregated into group mean scores to compare intervention and active comparator groups on this outcome.
Zarit Burden Scale, 12-item short form | 12 months
  This measure will be used to determine severity of caregiving-related burden among family caregivers who enroll in the study.This measure yields a score for each individual based on self-reports by family caregivers on the degree of caregiving impact on emotional, physical, social, and financial aspects of life. Individual scores will be aggregated into group mean scores to compare intervention and active comparator groups on this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Richard H Fortinsky, PhD, Principal Investigator — UConn Health
Locations (1):
- UConn Center on Aging, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levine AMP, Emonds EE, Smith MA, Rickles NM, Kuchel GA, Steffens DC, Ohlheiser A, Fortinsky RH. Pharmacist Identification of Medication Therapy Problems Involving Cognition Among Older Adults Followed by a Home-Based Care Team. Drugs Aging. 2021 Feb;38(2):157-168. doi: 10.1007/s40266-020-00821-7. Epub 2020 Dec 23. PMID 33354755
- [Derived] Fortinsky RH, Kuchel GA, Steffens DC, Grady J, Smith M, Robison JT. Clinical trial testing in-home multidisciplinary care management for older adults with cognitive vulnerability: Rationale and study design. Contemp Clin Trials. 2020 May;92:105992. doi: 10.1016/j.cct.2020.105992. Epub 2020 Mar 16. PMID 32194252